CLINICAL TRIAL: NCT01601522
Title: Peanut Allergy Oral Immunotherapy Desensitization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: AllerGen NCE Inc. (Industry); McMaster University (Other)
Responsible Party: Principal Investigator, Dr. Susan Waserman, Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB 07-348
Record Dates: First submitted 2011-07-27; First posted 2012-05-18 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — Histamine Antagonists; desloratadine; Ranitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oral Immunotherapy with placebo antihistamines (Experimental): 500 mg Peanut Protein with placebo antihistamines
  Interventions: Procedure: Peanut protein
- Double Placebo (Placebo Comparator): Placebo (Oat flour) and placebo antihistamines
  Interventions: Procedure: Oat flour
- Oral Immunotherapy with H1 and H2 antihistamines (Active Comparator): 500 mg Peanut Protein with Dosage of desloratidine 5 ml po od (0.5mg/ml = 2.5 mg) and ranitidine be 5ml (15mg/ml=75 mg) po bid.
  Interventions: Procedure: Peanut protein; Drug: Antihistamine

INTERVENTIONS:
Procedure: Peanut protein — 500 mg
  Other Names: Old Birginia Byrd Mill 12% Lightly Roasted Peanut Flour
  Arms: Oral Immunotherapy with H1 and H2 antihistamines; Oral Immunotherapy with placebo antihistamines
Procedure: Oat flour — 500 mg Oat flour
  Arms: Double Placebo
Drug: Antihistamine — Desloratidine 5 ml po od (0.5mg/ml = 2.5 mg) Ranitidine 5ml (15mg/ml=75 mg) po bid
  Other Names: Desloratadine and Ranitidine
  Arms: Oral Immunotherapy with H1 and H2 antihistamines

SUMMARY:
The purpose of the study is to determine how a type of treatment for peanut allergy known as oral desensitization works in the immune system.

Objectives

1. To determine whether premedication with desloratidine and ranitidine results in fewer side effects during desensitization procedure.
2. To assess quality of life in peanut allergic subjects before and after desensitization.
3. To compare serum metabolites in peanut allergic and non peanut allergic subjects.

DETAILED DESCRIPTION:
Allergic reactions to peanuts and tree nuts account for the majority of fatal and near fatal food allergic reactions, and the only treatment is complete avoidance of peanut. Despite avoidance, the majority of peanut allergic people will accidently ingest peanut. OIT has been shown to desensitize peanut allergic subjects (Hofmann et al. 2009). This would protect patients who have no other treatment, and may even form the basis for true tolerance to peanut in the future.

Objectives:

1. To determine whether premedication with desloratidine and ranitidine results in fewer side effects during desensitization procedure.
2. To assess quality of life in peanut allergic subjects before and after desensitization.
3. To compare serum metabolites in peanut allergic and non peanut allergic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 5 and 10 years of age.
* Patients will be confirmed to have peanut allergy based on a history of significant clinical symptoms within 60 minutes after the ingestion of peanut,the presence of specific IgE to peanut (a positive skin prick test to peanut, defined as a wheal 3 mm larger than that of the saline control; and a positive in vitro IgE [CAP-FEIA] result of >15 kU/L..
* Patients will also be accepted into the study if they have a clinical reaction to peanut ingestion within the past 6 months, a positive skin prick test to peanut as defined previously, and an in vitro peanut IgE (CAP-FEIA) result of 7 kU/L or greater.
* Subjects must be free of any clinically significant disease which may interfere with study evaluations.

Exclusion Criteria:

* Use of antihistamines or decongestant therapy 7 days prior to the clinic visit. (antihistamines eg. diphenhydramine, desloratadine etc or throughout the desensitization phase of the study.
* Patients who had an acute allergic reaction to food other than peanut, drugs, or stinging insects one month prior to the recruitment clinic visit
* Patients who have had a respiratory infection one month prior to the recruitment clinic visit.
* Patients with significant or uncontrolled asthma, (inhaled corticosteroids (fluticasone >500 mcg per day, ciclesonide >400 mcg per day or budesonide >800 mcg per day or the corresponding combination inhalers, oral prednisone in the preceding 1 month and FEV1 < 80% predicted). Nasal steroids, bronchodilators and leukotriene inhibitors will be permitted. If Prednisone is taken, it must also be stopped 1 month prior to blood being drawn if possible.
* Patients who received allergy injections (immunotherapy) to environmental allergens at any time in the past. Symptomatic atopic dermatitis or chronic urticaria which may interfere with ability to evaluate oral immunotherapy and /or requiring daily medication including antihistamines.
* Patients with problems related to compliance or following study instructions. Inability to come to hospital every 2 weeks for dose escalation.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2012-02; Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Adverse effects | 6-12 months
  Frequency and risk of adverse events, overall and stratified by organ system and severity

SECONDARY OUTCOMES:
Health related quality of life pre and post intervention | 6-12 months
  Pre and post OIT.
Eliciting doses to oral food challenge | 6-12 months
  Patients will be challenged at the end of the treatment period with peanut at the end to determine the change from threshold that they are able to tolerate.

OTHER OUTCOMES:
Immunological changes/Mechanistic outcomes | 6-12 months
  Various mechanistic outcomes/biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Susan Waserman, ME, Principal Investigator — McMaster University; Susan Waserman, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada